CLINICAL TRIAL: NCT02920736
Title: Value of Urine sTREM-1 on Early Predicting Secondary Acute Kidney Injury in Sepsis: a Mutilcenter and Prospective Clinical Study
Brief Title: Value of Urine sTREM-1 on Early Predicting AKI in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Chao Yang Hospital (Other); Peking University Shougang Hospital (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lixin Xie, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: shoufa2016-1-5015
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- sepsis with acute renal injury group: Based on definition of sepsis with Sepsis 3.0 and AKI was defined using KDIGO（Kidney Disease: Improving Global Outcomes） consensus definition of AKI.The group was the secondary AKI in sepsis patients
- sepsis non-acute renal injury group: The group was the non-AKI in sepsis patients
- control group: Approximately 110 persons(18-80years) with healthy physical examination and without liver and kidney dysfunction

SUMMARY:
The purpose of this study is to determine the value of urine sTREM-1 on early predicting secondary acute kidney injury in sepsis

DETAILED DESCRIPTION:
The clinical trial is a prospective, controlled study. All subjects were selected from among inpatients who were hospitalized between Sep.2016 and Dec.2018 in the Respiratory ICU, Surgical ICU and Emergency ICU of 6 general hospitals in Beijing. Based on the Sepsis 3.0,the population(500 subjects) selected met the diagnostic criteria. Based on the KDIGO (Nephrol Dial Transplant. 2012) defines AKI as 3 degrees, the subjects were divided into acute renal injury group (AKI group) and non-acute renal injury group (non-AKI group). Approximately 110 healthy volunteers enrolled as control group. Urine samples were collected from day 1 to day 28 in all patient groups (or to the terminal time point of death), serum samples were collected on days 1, 3, 5, 7, 10, and 14 and the samples were collected from healthy subjects on the day of enrollment. Blood was centrifuged at 3,000 rpm for 15 minutes, and urine at 2,000 rpm for 5 minutes. The supernatants were transferred to Eppendorf tubes and stored at -80°C. All the specimens were re-numbered before the experiment. Urine sTREM-1 was measured by a double antibody sandwich ELISA. This study was approved by the Ethics Committee of the CPLA General Hospital (project No.2014-113-02). The following clinical datas were recorded for all patients through the unified database software: (1) basic clinical information: hospital number, gender, age, underlying disease, hospital admission. (2) Daily vital signs after admission: body temperature, blood pressure, heart rate, respiratory rate, 24h urine volume, Glasgow score. (3) APACHE II score and SOFA score: arterial blood gas analysis, blood routine, C-reactive protein, procalcitonin, blood biochemistry (liver function, renal function, brain natriuretic peptide, blood electrolytes) The APACHE II score and the SOFA score were calculated. (4) 28-day outcome (survival or death). Statistical analyses were conducted by SPSS 16.0 (SPSS, Chicago,IL, USA) and a two-tailed P < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

All subjects meet the standards of sepsis 3.0 diagnostic criteria for the diagnosis of sepsis.

Exclusion Criteria:

The following situations can not occur when all subjects are enrolled

1. Age> 80 years or <18 years
2. Chronic renal insufficiency, renal transplantation
3. Blood purification treatment
4. AKI has occurred

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between Sep.2016 and Dec.2018 in the Respiratory ICU, Surgical ICU and Emergency ICU of 6 general hospitals in Beijing.All subjects were diagnosed with sepsis, based on the Sepsis 3.0.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
urine soluble triggering receptor expressed on myeloid cells-1 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: lixin xie, Ph.D., Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Ad-hoc working group of ERBP; Fliser D, Laville M, Covic A, Fouque D, Vanholder R, Juillard L, Van Biesen W. A European Renal Best Practice (ERBP) position statement on the Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guidelines on acute kidney injury: part 1: definitions, conservative management and contrast-induced nephropathy. Nephrol Dial Transplant. 2012 Dec;27(12):4263-72. doi: 10.1093/ndt/gfs375. Epub 2012 Oct 8. No abstract available. PMID 23045432